CLINICAL TRIAL: NCT02039700
Title: A Phase 1, Open-Label Study to Assess the Absolute Bioavailability of a Single Oral Dose of Lesinurad With Respect to an Intravenous Micro Tracer Dose of [14C]Lesinurad in Healthy Adult Male Subjects
Brief Title: Bioavailability of Lesinurad and Intravenous [14C]Lesinurad
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA594-131
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — lesinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lesinurad and [14C]lesinurad (Experimental): Single oral dose of lesinurad and single infusion of [14C]lesinurad
  Interventions: Drug: Lesinurad 400 mg; Drug: [14C]lesinurad (100 μg per 10 mL)

INTERVENTIONS:
Drug: Lesinurad 400 mg
Drug: [14C]lesinurad (100 μg per 10 mL)

SUMMARY:
This study will assess the absolute bioavailability of a single oral dose of lesinurad and evaluate the pharmacokinetic (PK) parameters of lesinurad and [14C]lesinurad in healthy adult male subjects.

DETAILED DESCRIPTION:
In this study a single dose of lesinurad will be administered after an overnight fast followed by a single 15-minute infusion of a radiolabeled intravenous micro tracer dose of [14C]lesinurad to assess the in vivo performance of lesinurad.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body weight ≥ 50 kg (110 lbs) and body mass index ≥ 18 and ≤ 30 kg/m2.
* Subject is free of any clinically significant disease or medical condition, per the Investigator's judgment

Exclusion Criteria:

* Subject has a history or suspicion of kidney stones.
* Subject has undergone major surgery within 3 months prior to Screening.
* Subject donated blood or experienced significant blood loss (>450 mL) within 12 weeks prior to Screening or gave a plasma donation within 4 weeks prior to Screening.
* Subject has inadequate venous access or unsuitable veins for repeated venipuncture.
* Subject does not have a normal or clinically acceptable physical examination, per the Investigator's judgment.
* Subject has clinically relevant abnormalities in blood pressure, heart rate, or body temperature, per the Investigator's judgment.
* Subject has Screening clinical safety laboratory parameters (serum chemistry, hematology, or urinalysis) that are outside the normal limits and are considered clinically significant by the Investigator.
* Subject has clinically relevant abnormalities in 12-lead electrocardiogram, per the Investigator's judgment.
* Subject has a Screening serum urate level > 7 mg/dL.
* Subject had radiation exposure that exceeds 5 mSv in the last 12 months or 10 mSv in the last 5 years. This includes radiation exposure from the present study or other clinical studies, including diagnostic X-rays and other medical exposures but excluding exposure to background radiation. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Characteristics of bioavailability in terms of lesinurad Pharmacokinetics (PK) profile from plasma. | Day 1 to Day 5
  PK profile in terms of maximum observed concentration (Cmax), time of occurrence of maximum observed concentration (Tmax), area under the concentration-time curve (AUC), apparent terminal half-life (t½), mean residence time (MRT), mean absorption time (MAT), and absolute bioavailability (F).
PK profile of [14C]lesinurad from plasma | Day 1 to Day 5
  PK profile in terms of Cmax, AUC, t½, MRT, total body clearance (CL), and volume of distribution at steady state (Vss).

SECONDARY OUTCOMES:
Incidence of Adverse Events and Changes in Laboratory, Electrocardiogram, and Vital Signs Parameters | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Madison, Wisconsin, United States